CLINICAL TRIAL: NCT02514759
Title: The Women's Clinic of Kansas City Teen Outreach Program Replication Study
Brief Title: Replication of the Teen Outreach Program in Kansas City
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philliber Research & Evaluation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Philliber10-15TWC
Record Dates: First submitted 2015-07-28; First posted 2015-08-04 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Teenage Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Teen Outreach Program (Experimental): TOP is a youth development and service learning program for youth designed to reduce teenage pregnancy and increase school success by helping youth develop a positive self-image, life management skills, and realistic goals. The TOP program model consists of three components implemented in school, after school, or in community settings over nine months: (1) weekly curriculum sessions, (2) community service learning, and (3) positive adult guidance and support. The TOP Changing Scenes Curriculum is separated into four age-/stage-appropriate levels, Level 1 is typically for youth ages 12 or 13 and Level 4 is typically for youth age 17. The intended program dosage for each participant is a minimum of 25 weekly sessions (one per week at 40-50 minutes each) and at least 20 hours of community service learning over nine months. One or two facilitators, who plan the order of sessions based on the needs and interest of youth, implemented TOP in a group of 10 to 25 youth.
  Interventions: Behavioral: The Teen Outreach Program
- Control group (No Intervention): The control group received business as usual.

INTERVENTIONS:
Behavioral: The Teen Outreach Program — Students received the Teen Outreach Program as described previously.
  Arms: The Teen Outreach Program

SUMMARY:
The Women's Clinic of Kansas City (TWC) replicated the Teen Outreach Program (TOP) across Kansas City, Missouri. The purpose of this study is to measure: one year after the end of the program year, what is TOP's impact on the treatment group's sexual activity and contraceptive use, relative to the control group, at one year following the program?

DETAILED DESCRIPTION:
TOP is a youth development and service learning program for youth ages 12 to 17 designed to reduce teenage pregnancy and increase school success by helping youth develop a positive self-image, life management skills, and realistic goals. The TOP program model consists of three components implemented in school, after school, or in community settings over nine months: (1) weekly curriculum sessions, (2) community service learning, and (3) positive adult guidance and support. The TOP Changing Scenes Curriculum is separated into four age-/stage-appropriate levels, Level 1 is typically for youth ages 12 or 13 and Level 4 is typically for youth age 17. The curriculum focuses on the presence of a consistent, caring adult; a supportive peer group; skill development; sexual health; and sexual behavior choices. The intended program dosage for each participant is a minimum of 25 weekly sessions (one per week at 40-50 minutes each) and at least 20 hours of community service learning over nine months. One or two facilitators, who plan the order of sessions based on the needs and interest of youth, implemented TOP in a group of 10 to 25 youth.

In this cluster randomized controlled trial, twelve of the highest-risk (based on highest teen births per zip code ranking in 2008) middle and high schools in the Kansas City Metropolitan Area were recruited to participate in the evaluation. After finalizing agreements with seven schools that agreed to participate, 7th- and 9th-grade teachers of core subjects (such as social studies and English) were recruited to participate. During the two years of sample enrollment, 21 teachers participated. At the start of each school year of sample enrollment, the study team assessed whether each participating teacher's class sections would be eligible for the evaluation based on the number of students enrolled (class sections were eligible if they had at least 10 students). Classes were

This study is a cluster randomized controlled trial across two cohorts. Stratification occurred at the teacher level; each teacher's classes were randomized to either TOP or the control condition. Random assignment occurred after acquiring parental consent and youth assent and administering the baseline survey. A passive consent process was used to notify parents that their youth would be participating in a youth development survey unless they opted out of the process. In addition, youth were given the option to not assent to any specific survey. Overall, youth in completed three surveys: (1) baseline, (2) 9-month post-baseline (immediate follow-up), and (3) 21-month post-baseline (1-year post-intervention follow-up). Students were surveyed in class using paper-and-pencil surveys; make-up surveys occurred during follow-up visits to the school over the final few weeks of school. Those chronically absent or no longer enrolled in the study schools were contacted via telephone to complete a telephone survey or via email to complete the survey online. Final efforts were made to visit youth who dropped out or who had been otherwise unreachable by going directly to their homes (if they still lived in the area); these youth were given a paper-and-pencil survey to complete. Students received a modest incentive for completing each survey.

ELIGIBILITY:
Inclusion Criteria:

* Has parental consent and student assent
* Attends one of the schools and/or classes chosen for the program

Exclusion Criteria:

* Lack of consent or assent

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1885 (Actual)
Dates: Start 2012-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Sexual activity | One year after the program (21 months)
  TOP's impact on the treatment group's sexual activity, relative to the control group, as measured by the questions "have you ever had sex" and "have you had sexual intercourse in the past three months".
Contraceptive use | One year after the program (21 months)
  TOP's impact on the treatment group's contraception use, relative to the control group, as measured by the question "have you had sexual intercourse in the past three months without using any method of birth control" and "have you had sexual intercourse in the past three months without using a condom".

SECONDARY OUTCOMES:
Grades | One year after the program (21 months)
  TOP's impact on the treatment group's course failures, relative to the control group, as measured by the question "Have you failed any courses for the whole year".
School suspensions | One year after the program (21 months)
  TOP's impact on the treatment group's school suspensions, relative to the control group, as measured by the question "in this past year have you been suspended from school".

CONTACTS AND LOCATIONS:
Overall Officials: Susan Philliber, PhD, Principal Investigator — Philliber Research Associates